CLINICAL TRIAL: NCT04555291
Title: Analgesic Efficiency of the Type 3 Quadratum Lumborum Block in Patients Undergoing Total Hip Arthroplasty : a Randomized Double Blinded Trial
Brief Title: Analgesic Effect of the QLB-3 for Patients Undergoing a Total Hip Surgery
Acronym: QLB-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-PP-13
Record Dates: First submitted 2020-08-11; First posted 2020-09-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Ropivacaïne 2 mg/ml (Experimental): Realization of the quadratum lumborum block type 3, ultrasounds' guided by the injection of 20 ml of ropivacaïne 2 mg/ml
  Interventions: Drug: Ropivacaine injection
- NACL (Placebo Comparator): Realization of the quadratum lumborum block type 3, ultrasounds' guided by the injection of 20 ml of NACL
  Interventions: Other: NACL

INTERVENTIONS:
Drug: Ropivacaine injection — Realization of the quadratum lumborum block type 3, ultrasounds' guided by the injection of 20 ml of ropivacaïne 2 mg/ml
  Arms: Drug Ropivacaïne 2 mg/ml
Other: NACL — Realization of the quadratum lumborum block type 3, ultrasounds' guided by the injection of 20 ml of NACL
  Arms: NACL

SUMMARY:
Total hip arthroplasty (THA) is one of the main elective orthopedic surgery. Recent studies have proven that patients undergoing an elective THA who are part of a fast track surgery program including an opioid free anesthesia (OFA) presented a decrease of mortality and a reduced in-hospital length of stay. Based on the anatomical knowledges, the Quadratus Lumborum Block seems to be an interesting locoregional technique for patients undergoing THA. So far, there is no recommanded locoregional aesthesia in this indication. The investigators hypothezised that QLB would give an efficient analgesia in the 24h following a THA.

Therefor, the study performed a prospective, randomized, double blind trial in the Nice Universitary hospital of Pasteur 2 and in Arnault Tzanck Institute among all patients who underwent THA, comparing a QLB using ropivacaïne 2mg/ml 20ml vs isotonic saline solution 20 ml.The main end-point is the decrease opiod consumption in the 24h following THA.

ELIGIBILITY:
Inclusion Criteria:

• All adult patients with unilateral programmed total hip prosthesis surgery are included in the absence of inclusion criteria.

* Obligation for all patients to be affiliated with social security
* Patient Informed Consent Signature

Exclusion Criteria:

* chronic opiod consumption
* pregnancy
* mental disorder that prevents the usage of the numeric analog scale
* Contra indications of the realization of QLB

  * Local infection
  * Allergic to the local anesthesia
  * Hemostasis disorder
  * Incapacity of giving the consent : individuals under guardianship by court order, or under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-10-06 (Estimated)

PRIMARY OUTCOMES:
Opoïd consumption | At 24 Hours
  The main end point of this study is the decrease of opiod consumption in the 24h following THA.

SECONDARY OUTCOMES:
morphine equivalent dose | At 48 Hours
  following surgery at rest and in motion

CONTACTS AND LOCATIONS:
Overall Officials: Rozier Romain, Principal Investigator — Anesthésie Réanimation - CHU de Nice
Locations (2):
- France (2):
  - CHU de nice - Anesthésie Réanimation, Nice, Alpes-Maritimes
  - Institut Arnaut Tzanck, Nice, Alpes-Maritimes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rozier R, Loiseleur A, Ciais C, Moulin O, Alais B, Marguerite K, Badia E, Tran L, Balbo J, Maurice-Szamburski A. Anterior quadratus lumborum block in total hip arthroplasty: a two-center, randomized, placebo-controlled trial showing no additional benefit over multimodal analgesia. Reg Anesth Pain Med. 2025 Feb 10:rapm-2024-106247. doi: 10.1136/rapm-2024-106247. Online ahead of print. PMID 39929638